CLINICAL TRIAL: NCT04455386
Title: Comparative Study on Accuracy of Different Diagnostic Methods of Lateral Ligament Complex Injury of Ankle
Brief Title: Diagnostic Study of Lateral Ligament Complex Injury of Ankle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Guo Qinwei, associated professor, Peking University Third Hospital
Other Study IDs: PKU-GUO-02
Record Dates: First submitted 2020-06-27; First posted 2020-07-02 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Chronic Instability of Ankle Joint; Lateral Ligament Complex Injury of Ankle
Keywords: Lateral Ligament complex; Ankle; Diagnostic Methods; Chronic Lateral Instability of Ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- stable: The anterior drawer test and/or talar tilt test are negative and the ankle joint is stable.
  Interventions: Diagnostic Test: Stress radiography,Anterior drawer test,Stress ultrasound,Computed tomography, Magnetic resonance imaging,Arthroscopy
- slightly instable: The anterior drawer test and/or talar tilt test are slightly positive and the ankle joint is partially instable.
  Interventions: Diagnostic Test: Stress radiography,Anterior drawer test,Stress ultrasound,Computed tomography, Magnetic resonance imaging,Arthroscopy
- obviously instable: The anterior drawer test and/or talar tilt test is significantly positive, with significantly instable. The ankle joint is completely instable and can featured with dimple sign.
  Interventions: Diagnostic Test: Stress radiography,Anterior drawer test,Stress ultrasound,Computed tomography, Magnetic resonance imaging,Arthroscopy

INTERVENTIONS:
Diagnostic Test: Stress radiography,Anterior drawer test,Stress ultrasound,Computed tomography, Magnetic resonance imaging,Arthroscopy — All patients suspected chronic ankle instability, will perform an anterior drawer test, stress ultrasound, computed tomography, magnetic resonance imaging of ankle. Patients with chronic ankle instability will be recommended to perform an arthroscopic repair if non-operative treatment failed.

SUMMARY:
Comparative Study on Accuracy of Different Diagnostic Methods of Lateral Collateral Ligament Injury of Ankle

DETAILED DESCRIPTION:
Background: The lateral ligament complex of ankle joint consisting of the anterior talofibular ligament (ATFL), the calcaneofibular ligament (CFL), and the posterior talofibular ligament (PTFL), is often injured by an ankle sprain. Improper diagnosis and treatment of lateral ligament complex injury are not only prone to recurrent sprain, pain, swelling and other symptoms, but also can lead to chronic lateral ankle instability, and osteoarthritis, which could seriously affect the joint motor function.

Method and objective: This study is a prospective diagnostic test. By comparing the sensitivity and specificity of stress X-ray, B-ultrasound, Computed tomography (CT), and Magnetic resonance imaging (MRI), and analyzing the imaging manifestations and characteristics of different diagnostic methods of lateral chronic ankle instability, We aim to propose the criteria of the imaging diagnosis of lateral ankle ligament injury.

ELIGIBILITY:
Inclusion Criteria:

* Chronic lateral ankle ligament injury due to ankle sprain in patients over 16 years of age.

Exclusion Criteria:

* Acute and subacute injury of the lateral ligament complex of the ankle joint (less than 3 months), malalignment of ankle (more than 5 degrees), osteoarthritis (stage IV).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic lateral ligament complex injury of the ankle were divided into 3 groups and each group with 25 cases, according to the anterior drawer test and talar tilt test.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
anterior talar translation and talar tilt | before operation
  Assess the instability through stress X ray of the ankle
length of ATFL and CFL in relax and stress position | before operation
  Assess the instability through Ultrasound of the ankle
Morphology of ATFL and CFL | before operation
  Assess the ATFL and CFL through MRI of the ankle
status of ATFL and CFL | during operation
  evaluation of ATFL and CFL during operation

SECONDARY OUTCOMES:
avulsion fracture | before operation
  avulsion fracture found by X ray, Ultrasound, CT or MRI
osteophyte | before operation
  osteophyte found by X ray, Ultrasound, CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No